CLINICAL TRIAL: NCT00716339
Title: Pseudophakic Accommodation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: EK 481/2004
Record Dates: First submitted 2008-07-09; First posted 2008-07-16 (Estimated); Last update posted 2008-07-16 (Estimated); Status verified 2008-07

CONDITIONS: Cataract
Keywords: pseudophakic accommodation
MeSH Terms: conditions — Cataract | interventions — Information Motivation Behavioral Skills Model

ARMS (2):
- 1 (Active Comparator): motivated
  Interventions: Behavioral: motivation
- 2 (No Intervention): control

INTERVENTIONS:
Behavioral: motivation
  Arms: 1

SUMMARY:
Purpose:

The aim of this study was to compare the effect of ciliary body training as proposed by manufacturers of accommodating IOLs and patient motivation on the pseudoaccommodative ability with a standard intraocular lens (SA60AT).

Setting:

Department of Ophthalmology, Medical University of Vienna.

Methods:

This randomized, controlled, examiner-masked study comprised 80 eyes of 40 patients that underwent standard cataract surgery. Patients were randomly assigned to a "motivated" or "non-motivated" (control) group. In the motivated group, subjects were told to take part in a special protocol to improve their near-reading ability after cataract surgery and were instructed not to use near adds for at least 3 months. Follow-up examinations included best-corrected distance visual acuity (VA), distance-corrected near VA, best-corrected near VA, defocus curve and reading speed, as well as pilocarpine-, cyclopentolate- and nearpoint-induced IOL shift assessed with partial coherence interferometry.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from age-related cataract who are enrolled for cataract surgery.
* Age 50 to 75 years
* < 1 D of corneal astigmatism, estimated postoperative VA of 20/30 or better and IOL power between 16 and 27 dpt

Exclusion Criteria:

* Patients with complications during cataract surgery or during the postoperative period, significant other ophthalmic diseases such as glaucoma, diabetic retinopathy, etc., or ophthalmic surgery other than cataract surgery

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40

PRIMARY OUTCOMES:
visual acuity (best-corrected distance VA, distance-corrected near VA, best-corrected near VA)

SECONDARY OUTCOMES:
IOL shift (pilocarpine-, cyclopentolate- and nearpoint-induced) assessed with partial coherence interferometry

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Vienna, Department of Ophthalmology, Vienna, Vienna, Austria